CLINICAL TRIAL: NCT01789164
Title: Measure of Cerebrovascular Dysfunction After Truamatic Brain Injury With Functional Near Infrared Spectroscopy
Brief Title: Measure of Cerebrovascular Dysfunction After TBI With fNIRS
Status: Completed | Type: Observational
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ramon Diaz-Arrastia, Director of Clinical Research, Uniformed Services University of the Health Sciences
Other Study IDs: G189AP-S2
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Traumatic Brain Injury; Post-concussion Syndrome
Keywords: TBI; fNIRS; hypercapnea; Cerebrovascular reactivity
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Concussion Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy group: Healthy group with no history of TBI or concussion. Gender matched non-TBI volunteers
- TBI group: Males and females between 18 and 60 years who have a diagnosis of TBI and are symptomatic with DSM-IV Research Criteria for Post-Concussional Disorder (see below), gender matched non-TBI volunteers

SUMMARY:
The goal of this project is to determine if it is possible to assess Cerebrovascular Reactivity (CVR) to hypercapnia with functional Near Infrared Spectroscopy (fNIRS). Such a method would be particularly helpful in traumatic brain injury (TBI), where objective measures are needed, and would greatly expand the capacity to make such assessments in standard clinical practice.

DETAILED DESCRIPTION:
The prospective study design will consist of two study groups; the experimental group and the control group. In the Experimental Group (Group 1) we will enroll adult participants with TBI with persistent post-concussion symptoms or abnormalities on neuropsychological testing. In Group 2 we will enroll adult participants to serve as age and gender-matched healthy controls. Our goal is to recruit 100 subjects total in two groups of age and gender matched subjects, as follows: TBI (n = 50) and non-TBI (n = 50).

Participants in both groups will undergo NIRS testing with hypercapnia challenge, to measure the increase in hemodynamic flow signal during hypercapnia challenge via 2 methods, the breath holding and the Douglas bag methods. We will test intersessional validity of the NIRS-hypercapnia challenge in the first 20 (10 TBI and 10 non-TBI) subjects who are willing to return for a second visit of repeat testing.

The NIRS system is composed of 4 light sources and 10 detectors with a 16 point configuration system applied on the forehead of the subject. In our experiment, light intensity collected at each detector will be transformed into a signal related to the local concentrations of oxy- and de-oxyhemoglobin during the challenge. Each experiment will give a set of subject data, consisting of the peak amplitude and time-to-peak of the hemodynamic signals measured.

ELIGIBILITY:
Inclusion Criteria:

1. ALL participants (TBI and non-TBI) subjects Males and females, ages 18 to 60 years, inclusive Able to read, write, speak and understand English
2. A history of TBI
3. Persistent post-concussive symptoms, according to the DSM-IV Research
4. Criteria for Post-Concussional Disorder, including:

   * Evidence from neuropsychological testing of difficulty in attention or memory. (refers to neuropsychological testing done as a part of the patient's hospital or rehabilitation care not as a part of screening for this study)
   * Three or more of the following symptoms, which started shortly after the trauma and persist for at least three months:

     * Fatigability
     * Disordered sleep
     * Headache
     * Vertigo or dizziness
     * Irritability or aggression
     * Anxiety, depression, or affective instability
     * Changes in personality (e.g. social or sexual inappropriateness)
     * Apathy or lack of spontaneity

Symptoms in criteria (a) and (b) must have their onset after trauma, or there was a significant worsening of pre-existing symptoms after trauma.

Exclusion Criteria:

1. History or evidence of pre-existing neurological or psychiatric disorder not related to TBI, such as:

   * Multiple sclerosis, pre- or co-existing
   * Stroke (other than stroke at the time of TBI)
   * Pre-existing developmental disorder
   * Pre-existing epilepsy
   * Pre-existing major depressive disorder
   * Pre-existing schizophrenia
2. Known allergy to latex (used in the NIRS apparatus band applied to the forehead)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Males and females (military health care beneficiaries and non military health care beneficiaries) between 18 and 60 years who have a diagnosis of TBI and are symptomatic with DSM-IV Research Criteria for Post-Concussional Disorder (see below), gender matched non-TBI volunteers.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reproducibility of CVR measurements with fNIRS during intersession and intra-session testing | Two years
  Establish reproducibility of CVR measurements with fNIRS during intersession and intra-session testing. Additionally, we will examine two methods of producing hypercapnia, breath holding and the Douglas bag methods to establish whether the two methods give similar NIRS results.

SECONDARY OUTCOMES:
Examine the following hypothesis: TBI subjects have a lower CVR compared to healthy controls | Two years

OTHER OUTCOMES:
The degree of CVR disruption correlates with the severity of TBI or post-concussive symptoms | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Diaz-Arrastia, MD, PhD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Center for Neuroscience and Regenerative Medicine (CNRM), Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kenney K, Amyot F, Haber M, Pronger A, Bogoslovsky T, Moore C, Diaz-Arrastia R. Cerebral Vascular Injury in Traumatic Brain Injury. Exp Neurol. 2016 Jan;275 Pt 3:353-366. doi: 10.1016/j.expneurol.2015.05.019. Epub 2015 Jun 3. PMID 26048614
- [Result] Amyot F, Kenney K, Spessert E, Moore C, Haber M, Silverman E, Gandjbakhche A, Diaz-Arrastia R. Assessment of cerebrovascular dysfunction after traumatic brain injury with fMRI and fNIRS. Neuroimage Clin. 2020;25:102086. doi: 10.1016/j.nicl.2019.102086. Epub 2019 Nov 11. PMID 31790877
- [Derived] Reddy P, Izzetoglu M, Shewokis PA, Sangobowale M, Diaz-Arrastia R, Izzetoglu K. Evaluation of fNIRS signal components elicited by cognitive and hypercapnic stimuli. Sci Rep. 2021 Dec 6;11(1):23457. doi: 10.1038/s41598-021-02076-7. PMID 34873185